CLINICAL TRIAL: NCT01626976
Title: A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo Controlled, Single Dose Escalating Study To Assess The Safety, Tolerability And Pharmacokinetics Of PF-06282999 Administered Orally In Healthy Adult Subjects
Brief Title: A Study To Assess The Safety, Tolerability And Pharmacokinetics Of PF-06282999 Administered Orally In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5211001
Record Dates: First submitted 2012-05-30; First posted 2012-06-25 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics; oral; single ascending dose; placebo-controlled; healthy subjects
MeSH Terms: interventions — 2-(6-(5-chloro-2-methoxyphenyl)-4-oxo-2-thioxo-3,4-dihydropyrimidin-1(2H)-yl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Cohort 3 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Cohort 4 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo
- Cohort 5 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo

INTERVENTIONS:
Drug: PF-06282999 — Solution, doses range from 20 to 200 mg, single dose
  Arms: Cohort 1
Drug: Placebo — Solution, single dose
  Arms: Cohort 1
Drug: PF-06282999 — Methylcellulose suspension, doses range 125 to 500 mg, single dose
  Arms: Cohort 2
Drug: Placebo — suspension, single dose
  Arms: Cohort 2
Drug: PF-06282999 — Methylcellulose or simethicone suspension, doses range 200 to 500 mg, single dose
  Arms: Cohort 3
Drug: Placebo — suspension, single dose
  Arms: Cohort 3
Drug: PF-06282999 — Methylcellulose or simethicone suspension, 500 mg dose, single dose
  Arms: Cohort 4
Drug: Placebo — suspension, single dose
  Arms: Cohort 4
Drug: PF-06282999 — Simethicone or methylcellulose suspension, up to 1500 mg, single dose
  Arms: Cohort 5
Drug: Placebo — suspension, single dose
  Arms: Cohort 5

SUMMARY:
This is the first-in-human study for an oral investigational compound, PF-06282999, in order to assess its safety, tolerability and pharmacokinetics in humans across a wide range of dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Women must be of non-childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including clinically significant drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf] | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Area Under the Curve From Time Zero to 24 hour [AUC24] | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours post-dose
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Apparent Oral Clearance (CL/F) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Apparent Volume of Distribution (Vz/F) | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose
Amount of Unchanged Drug Excretion in Urine from Zero to 24 hours (Ae24) | 0 to 24 hours post-dose
Percent of Dose Excreted in Urine as Unchanged Drug from Zero to 24 hours (Ae24%) | 0 to 24 hours post-dose
Renal Clearance (CLr) | 0 to 24 hours post-dose
Oral temperature | 0, 1, 2, 4, 8, 12,16, 24, 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5211001&StudyName=A%20Study%20To%20Assess%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20PF-06282999%20Administered%20Orally%20In%20Healthy%20Adult%20Subjects